CLINICAL TRIAL: NCT02875743
Title: Incidence of Invasive Fungal Disease in Patients Receiving Immunosuppressive Therapy, Intensive Chemotherapy or Reduced Intensity Haematopoietic Stem Cell Transplantation on Posaconazole Prophylaxis
Brief Title: King's Invasive Aspergillosis Study II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KIASII
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Aplastic Anemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Bone Marrow Transplantation
MeSH Terms: conditions — Anemia, Aplastic; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole (Experimental)
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole

SUMMARY:
Invasive fungal disease (IFD) is an important cause of mortality and morbidity in patients undergoing intensive chemotherapy or transplantation.

This current study aims to assess the impact of prophylactically using the broad-spectrum anti-fungal agent posaconazole on the incidence of IFD in high risk patients with aplastic anaemia and those undergoing intensive chemotherapy, for example for acute myeloid leukaemia, and allogeneic stem cell transplantation.

ELIGIBILITY:
INCLUSION CRITERIA

1. Adult ≥ 18 years
2. Patients with aplastic anaemia, MDS or AML undergoing: IST; or Intensive chemotherapy such as induction chemotherapy; or RIC allogeneic HSCT
3. Able to swallow and retain orally administered medication

EXCLUSION CRITERIA

1. Refusal or inability to consent
2. Autologous HSCT
3. Contraindicated medications
4. Current evidence of IFD diagnosis or treatment
5. Enrolled in another study requiring alternative antifungal prophylaxis or treatment
6. Women who are pregnant or lactating
7. Women who are unable to use and apply with effective contraception without interruption throughout the duration of study drug therapy and not willing to have further pregnancy tests during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of IFD in all treatment groups (aplastic anaemia with IST, chemotherapy only, RIC allograft) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom